CLINICAL TRIAL: NCT04657094
Title: A Phase 2 Trial of Acalabrutinib for the Treatment of Relapsed/Refractory Autoimmune Hemolytic Anemia
Brief Title: Acalabrutinib for the Treatment of Relapsed or Refractory Autoimmune Hemolytic Anemia in Patients With Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20311; NCI-2020-10529 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20311 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Autoimmune Hemolytic Anemia; Chronic Lymphocytic Leukemia; Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Warm Antibody Autoimmune Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (acalabrutinib) (Experimental): Patients receive acalabrutinib PO BID on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Treatment with acalabrutinib may be continued beyond 12 cycles for a maximum of 36 cycles if, in the opinion of the treating physician, the patient might benefit from ongoing therapy.
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP-196; Bruton Tyrosine Kinase Inhibitor ACP-196; Calquence

SUMMARY:
This phase II trial studies the effect of acalabrutinib in treating autoimmune hemolytic anemia that has come back (relapsed) or has not responded to previous treatment (refractory) in patients with chronic lymphocytic leukemia. Acalabrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the efficacy of acalabrutinib in chronic lymphocytic leukemia (CLL) patients with relapsed or refractory autoimmune hemolytic anemia (AIHA).

SECONDARY OBJECTIVES:

I. Evaluate acalabrutinib's ability to induce short term and sustained hemoglobin response.

II. Assess the toxicity of acalabrutinib. III. Evaluate efficacy of acalabrutinib in CLL.

EXPLORATORY OBJECTIVE:

I. Assess the effect of acalabrutinib on T-cell functionality in an autoimmune disorder.

OUTLINE:

Patients receive acalabrutinib orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Treatment with acalabrutinib may be continued beyond 12 cycles for a maximum of 36 cycles if, in the opinion of the treating physician, the patient might benefit from ongoing therapy.

After completion of study treatment, patients are followed up at 30 days and at least every 4 months for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Eastern Cooperative Oncology Group (ECOG) =< 2
* "Warm" or "cold" AIHA in patients with CLL, relapsed/refractory (RR) after first line treatment with oral prednisone (with or without rituximab), defined as:

  * Anemia (hemoglobin [Hgb] =< 10 g/dL; or Hgb > 10 g/dL dependent on transfusions or maintenance therapy (rituximab, cyclosporin, etc) to maintain this level of hemoglobin, and
  * Laboratory evidence of hemolysis - presence of 3 of 4 markers (increased reticulocyte count, increased indirect bilirubin, increased lactate dehydrogenase, absent haptoglobin)
* Positive direct antiglobulin test (DAT) (score >= 1+) - either immunoglobulin G (IgG) DAT, C3 DAT, or both. Eligibility of patients with Coombs-negative AIHA should be confirmed by the trial investigator at each respective study site
* Histologically or flow cytometry confirmed diagnosis of CLL/small lymphocytic lymphoma (SLL)
* Participant must be able to swallow tablets or capsules
* Absolute neutrophil count (ANC) >= 500/mm^3 unless due to disease involvement in the bone marrow or autoimmune neutropenia (within 30 days prior to day 1 of protocol therapy)
* Platelets >= 30,000/mm^3 unless due to disease involvement in the bone marrow or autoimmune thrombocytopenia (Evans syndrome) (within 30 days prior to day 1 of protocol therapy)
* Direct bilirubin =< 3.0 x upper limit of normal (ULN) (within 30 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase (AST) =< 3.0 x ULN (within 30 days prior to day 1 of protocol therapy)
* Alanine aminotransferase (ALT) =< 3.0 x ULN (within 30 days prior to day 1 of protocol therapy)
* Creatinine clearance of >= 30 mL/min per 24 hour urine test or the Cockcroft-Gault formula (within 30 days prior to day 1 of protocol therapy)
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (prothrombin time [PT]) < 2 x ULN (within 30 days prior to day 1 of protocol therapy). If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants (within 30 days prior to day 1 of protocol therapy)
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) < 2 x ULN (within 30 days prior to day 1 of protocol therapy). If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants (within 30 days prior to day 1 of protocol therapy)
* Seronegative for human immunodeficiency virus (HIV) Ag/Ab combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative), and syphilis (rapid plasma reagin [RPR]) (within 30 days prior to day 1 of protocol therapy)

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test within the screening window prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females of childbearing potential to use highly effective methods of birth control or abstain from heterosexual activity starting with the first dose of study therapy through 2 days after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Therapeutic anticancer antibodies within 3 weeks
* Radio- or toxin-immunoconjugates within 10 weeks
* BH3-mimetic venetoclax, PI3K inhibitors and other "targeted" therapy- within 6 half-lives
* Ibrutinib, acalabrutinib or another BTK inhibitor within 12 months
* Patients on stable chronic AIHA treatments are allowed provided the dose has not changed in the 4 weeks prior to enrollment
* Allogeneic stem cell transplant within 1 year prior to day 1 of protocol therapy, or ongoing immunosuppressive therapy for chronic graft versus host disease (cGVHD)
* Chemotherapy, radiation therapy, biological therapy, immunotherapy within 21 days prior to day 1 of protocol therapy
* Strong CYP3A4 inducers/ inhibitors. If the patient requires a strong CYP3A inhibitor/inducer, they should not be enrolled even if it could be held for 14 days before the first dose of study drug
* Proton pump inhibitors (but patients who switch to H2-receptor antagonists or antacids are eligible for enrollment)
* Chronic use of corticosteroids (> 2 weeks) in excess of prednisone 60 mg/day or its equivalent within 4 weeks prior to start of study therapy. Rescue steroids are allowed during trial
* Vitamin K antagonists
* Known intolerance to acalabrutinib
* History of bleeding disorders or with active bleeding
* Patients with suspected or confirmed progressive multifocal leukoencephalopathy (PML)
* Patients with history of stroke or intracranial hemorrhage within 6 months
* Inadequate recovery from adverse events related to prior therapy to grade 1 or baseline (excluding grade 2 alopecia and neuropathy)
* Active uncontrolled infection
* Known history of immunodeficiency virus (HIV) infection

  * Subjects who have an undetectable or unquantifiable HIV viral load with CD4 > 300 and are on highly active antiretroviral therapy (HAART) medication are allowed. Testing to be done only in patients suspected of having infections or exposures
* Active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)

  * Participants who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Note that intravenous immunoglobulin therapy (IVIG) administration may lead to positive anti-HBc test result
  * Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded
* Major surgery (requiring general anesthesia) within 28 days prior to initiation of therapy
* Has difficulty with or is unable to swallow oral medication, or has significant gastrointestinal disease that would limit absorption of oral medication
* History of prior malignancy except:

  * Malignancy treated with curative intent and no known active disease present for >= 2 years prior to initiation of therapy on current study
  * Adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease
  * Adequately treated in situ carcinomas (e.g., breast, cervical, esophageal, etc.) without evidence of disease
  * Asymptomatic prostate cancer managed with "watch and wait" strategy
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or left ventricular ejection fraction (LVEF) =< 40%
* Psychiatric illness/social situations that would limit compliance with study requirements
* Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2026-02-27 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Danilov, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Acalabrutinib)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Acalabrutinib)
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 59 [53 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Autoimmune Hemolytic Anemia (AIHA) - Overall Response Rate (ORR)
Description: ORR is defined as proportion of patients who achieve complete response (CR) and partial response (PR). The probability of having AIHA-ORR at 6 cycles were measured and reported with 95% exact confidence interval (CI). An exact binomial test against a null hypothesis of 30% rate was performed at the 1-sided alpha of 0.05 to determine whether the AIHA-ORR rate at 6 cycles is disappointing or promising.
Time Frame: Participants were assessed at the end of the 6-week therapy.
Population: Among the 4 enrolled participants, one was in-evaluable for not finishing 6 cycles of the study treatment due to toxicity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Acalabrutinib)
Number analyzed (Participants) | 3
percentage of participants | 67 [9 to 99]

ADVERSE EVENTS:
Time Frame: From the initial study treatment up to 12 months after the end of the treatment, approximately two years.
Arm/Group | Treatment (Acalabrutinib)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Acalabrutinib) (N=4)
DRESS Syndrome (Immune system disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Acalabrutinib) (N=4)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Dental Fractures (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Neck Numbness (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
DRESS Syndrome (Immune system disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (3)
Lymphocyte count increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (6)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT04657094/Prot_SAP_000.pdf